CLINICAL TRIAL: NCT02603718
Title: An Applicative On-line EEG Tool for Enhancing Treatment Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reuth Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-3
Record Dates: First submitted 2015-10-14; First posted 2015-11-13 (Estimated); Last update posted 2019-09-13 (Actual); Status verified 2018-05

CONDITIONS: Stroke Rehabilitation
Keywords: Stroke; On-line EEG; BEI index; Attention; Rehabilitation
MeSH Terms: conditions — Stroke | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard physical therapy treatment with feedback (Experimental): Standard physical therapy rehabilitation is administered to stroke patients. Attention level of the patient gathered with an EEG tool is measured, and provided to both therapist and patient on-line during one of the two treatments.
  Interventions: Other: Rehabilitation treatment
- Standard physical therapy treatment without feedback (Experimental): Standard physical therapy rehabilitation is administered to stroke patients. Attention level of the patient gathered with an EEG tool is measured but feedback is not provided.
  Interventions: Other: Rehabilitation treatment

INTERVENTIONS:
Other: Rehabilitation treatment

SUMMARY:
The purpose of this study is to investigate the efficacy of a simple and easy to use tool that can extract relevant attention-related markers - Brain Engagement Index (BEI) from ongoing EEG. During standard rehabilitative physical therapy sessions.

DETAILED DESCRIPTION:
This research aims at assessing and fine tuning the effectiveness of a unique tool for online guidance of neural rehabilitation. The tool monitors patient attention level and guides the therapist online regarding the effectiveness of the current exercise employed. It is well established that maintaining a high level of attention plays a major role in the clinical outcome in rehabilitation. The monitoring is achieved using a cheap and simple to use EEG system and a breakthrough signal processing algorithm. The feedback provides the caregiver and patient with online information regarding the effectiveness of attention recruited during a given exercise. Furthermore, the investigators are developing and fine-tuning a set of guidelines to attain optimal attention levels. These guide lines include : Choosing an appropriate goal/movement for each patient; Regulating the optimal degree of effort by changing the difficulty level of the exercise, changing the exercise or suggesting a short rest period; Integrating supportive exercises such as stretches, strengthening of stabilizers normalization of muscle tone, sensory stimulation etc. which may enhance the performance of the target goal/movement; Motivating patients to exert more effort; And taking advantage of the quality control aspect of the BEI index in-order to augment attention of both therapist and patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients after stroke willing

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2017-08-28 (Actual); Study Completion 2017-08-28 (Actual)

PRIMARY OUTCOMES:
Clinical outcome on a -3 to +3 scale | Change in performance between pre & post treatment, will be assessed twice, in the feedback session and non-feedback session. Each participant will be assessed twice within two weeks from recruitment to the study.
  video
Mean brain engagement index during treatment. | During the whole treatment session, each participant will be assessed twice within two weeks from recruitment to the study.
  scale from zero to one, the time in which the measure excedes a predefined threshhold level during tretment
Session effectiveness index | Through treatment sessions, each participant will be assessed twice within two weeks from recruitment to the study.
  Scale from 1 to 3, the average of effectiveness evaluations for all the treatments in each session was used as the session effectiveness index

CONTACTS AND LOCATIONS:
Locations (1):
- Reuth Rehabilitation Hospital, Tel Aviv, Israel

REFERENCES:
- [Derived] Bartur G, Joubran K, Peleg-Shani S, Vatine JJ, Shahaf G. An EEG Tool for Monitoring Patient Engagement during Stroke Rehabilitation: A Feasibility Study. Biomed Res Int. 2017;2017:9071568. doi: 10.1155/2017/9071568. Epub 2017 Sep 24. PMID 29147661